CLINICAL TRIAL: NCT05818956
Title: A Randomized, Open-label, Single-dose, Three-way Crossover Evaluation of the Effect of Food on the Pharmacokinetics, Safety, and Tolerability of TAK-227 in Healthy Adult Participants
Brief Title: A Study of TAK-227 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-227-1001
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Sequence 1: (Treatment A + Treatment B + Treatment C) (Experimental): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 under fasting condition as Treatment A, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C. There will be a washout period of at least 4 days between each dosing.
  Interventions: Drug: TAK-227
- Sequence 2: (Treatment B + Treatment C + Treatment A) (Experimental): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 under fasting condition as Treatment A . There will be a washout period of at least 4 days between each dosing.
  Interventions: Drug: TAK-227
- Sequence 3: (Treatment C + Treatment A + Treatment B) (Experimental): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 under fasting condition as Treatment A, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B. There will be a washout period of at least 4 days between each dosing.
  Interventions: Drug: TAK-227
- Sequence 4: (Treatment A + Treatment C + Treatment B) (Experimental): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 under fasting condition as Treatment A, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B. There will be a washout period of at least 4 days between each dosing.
  Interventions: Drug: TAK-227
- Sequence 5: (Treatment B + Treatment A + Treatment C) (Experimental): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 under fasting condition as Treatment A, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C. There will be a washout period of at least 4 days between each dosing.
  Interventions: Drug: TAK-227
- Sequence 6: (Treatment C + Treatment B + Treatment A) (Experimental): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 under fasting condition as Treatment A. There will be a washout period of at least 4 days between each dosing.
  Interventions: Drug: TAK-227

INTERVENTIONS:
Drug: TAK-227 — TAK-227 capsules.

SUMMARY:
The main aim of this study is to test the effects of food consumption with sponsor compound TAK-227 in healthy participants. The study will also measure side effects, and to check how much TAK-227 stays in the blood over time to work out the best dose.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-227. This study will assess the effect of food on single-dose of TAK-227 in healthy participants.

The study will enroll approximately 24 participants. A single dose of 50 milligram (mg) TAK-227 will be administered orally under one of 3 different feeding conditions.

* Fasting (Treatment A),
* Fed following a high-fat or high-calorie meal prior to dosing (Treatment B), and
* Fed following a high-fat or high-calorie meal after dosing (Treatment C)

Participants will be randomly assigned to 1 of the 6 treatments sequences based on the 3 feeding conditions.

* Sequence 1: (Treatment A + Treatment B + Treatment C)
* Sequence 2: (Treatment B + Treatment C + Treatment A)
* Sequence 3: (Treatment C + Treatment A + Treatment B)
* Sequence 4: (Treatment A + Treatment C + Treatment B)
* Sequence 5: (Treatment B + Treatment A + Treatment C)
* Sequence 6: (Treatment C + Treatment B + Treatment A)

All participants will receive all 6 treatment regimens. This is a single-center trial. Participants will be followed up for up to 7 days after the last dose of study drug for a follow-up assessment. The overall time to participate in this study is approximately 40 days including screening period and follow-up period.

ELIGIBILITY:
Inclusion Criteria

Participants must fulfill the following inclusion criteria to be eligible for participation in the study:

* Body mass index (BMI) greater than or equal to (>=) 18 and less than or equal to (<=) 32.0 kilogram per square meter (kg/m^2) at screening visit.
* Continuous non-smoker who has not used nicotine and tobacco containing products for at least 3 months prior to the first dosing based on participant self-reporting.

Exclusion Criteria:

Participants must not be enrolled in the study if they meet any of the following criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* Drink alcohol in excess of 21 units per week for males or 14 units per week for females, with one unit equal to (=) 150 milliliter (mL) of wine or 360 mL of beer or 45 mL of 45 percent (%) alcohol.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
* Unable to refrain from or anticipates the use of:

  * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Medication listed as part of acceptable birth control methods will be allowed. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first study drug administration. Hormone replacement therapy will also be allowed.
  * Any drugs known to be significant inducers or inhibitors of Cytochrome P450 (CYP)3A4 enzymes and/or P-glycoprotein (gp), including St. John's Wort, within 28 days prior to the first dosing and throughout the study. Appropriate sources (example, Flockhart Table TM) will be consulted to confirm lack of pharmacokinetic (PK)/pharmacodynamics interaction with study drug.
  * Chronic use of non-steroidal anti-inflammatory (define as more that 7 days of use) within 2 weeks prior to screening and throughout the study.
* Donation of blood or significant blood loss within 56 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/7a014b6ccea84ef4?idFilter=%5B%22TAK-227-1001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at single investigative site in the United States from 25 May 2023 to 26 June 2023.
Pre-assignment Details: Healthy participants were randomized in each of the 6 treatment sequences of this 3-period cross over study to receive a 50 milligram (mg) capsule of TAK-227 in the fasting state (Treatment A), fed predose state following a high-fat/high-calorie meal 30 minutes prior to dosing (Treatment B), or fed postdose state following a high-fat/high-calorie meal 30 minutes after dosing (Treatment C).
Groups:
- Treatment Sequence 1: (Treatment A + Treatment B + Treatment C): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 under fasting condition as Treatment A, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C. There was a washout period of not less than 4 days between each treatment period.
- Treatment Sequence 2: (Treatment B + Treatment C + Treatment A): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 under fasting condition as Treatment A . There was a washout period of not less than 4 days between each treatment period.
- Treatment Sequence 3: (Treatment C + Treatment A + Treatment B): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 under fasting condition as Treatment A, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B. There was a washout period of not less than 4 days between each treatment period.
- Treatment Sequence 4: (Treatment A + Treatment C + Treatment B): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 under fasting condition as Treatment A, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B. There was a washout period of not less than 4 days between each treatment period.
- Treatment Sequence 5: (Treatment B + Treatment A + Treatment C): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 under fasting condition as Treatment A, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C. There will be a washout period of not less than 4 days between each treatment period.
- Treatment Sequence 6: (Treatment C + Treatment B + Treatment A): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 under fasting condition as Treatment A. There will be a washout period of not less than 4 days between each treatment period.
Period: Treatment Period 1 (2 Days)
Arm/Group | Treatment Sequence 1: (Treatment A + Treatment B + Treatment C) | Treatment Sequence 2: (Treatment B + Treatment C + Treatment A) | Treatment Sequence 3: (Treatment C + Treatment A + Treatment B) | Treatment Sequence 4: (Treatment A + Treatment C + Treatment B) | Treatment Sequence 5: (Treatment B + Treatment A + Treatment C) | Treatment Sequence 6: (Treatment C + Treatment B + Treatment A)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (4 Days)
Arm/Group | Treatment Sequence 1: (Treatment A + Treatment B + Treatment C) | Treatment Sequence 2: (Treatment B + Treatment C + Treatment A) | Treatment Sequence 3: (Treatment C + Treatment A + Treatment B) | Treatment Sequence 4: (Treatment A + Treatment C + Treatment B) | Treatment Sequence 5: (Treatment B + Treatment A + Treatment C) | Treatment Sequence 6: (Treatment C + Treatment B + Treatment A)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (2 Days)
Arm/Group | Treatment Sequence 1: (Treatment A + Treatment B + Treatment C) | Treatment Sequence 2: (Treatment B + Treatment C + Treatment A) | Treatment Sequence 3: (Treatment C + Treatment A + Treatment B) | Treatment Sequence 4: (Treatment A + Treatment C + Treatment B) | Treatment Sequence 5: (Treatment B + Treatment A + Treatment C) | Treatment Sequence 6: (Treatment C + Treatment B + Treatment A)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (4 Days)
Arm/Group | Treatment Sequence 1: (Treatment A + Treatment B + Treatment C) | Treatment Sequence 2: (Treatment B + Treatment C + Treatment A) | Treatment Sequence 3: (Treatment C + Treatment A + Treatment B) | Treatment Sequence 4: (Treatment A + Treatment C + Treatment B) | Treatment Sequence 5: (Treatment B + Treatment A + Treatment C) | Treatment Sequence 6: (Treatment C + Treatment B + Treatment A)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (2 Days)
Arm/Group | Treatment Sequence 1: (Treatment A + Treatment B + Treatment C) | Treatment Sequence 2: (Treatment B + Treatment C + Treatment A) | Treatment Sequence 3: (Treatment C + Treatment A + Treatment B) | Treatment Sequence 4: (Treatment A + Treatment C + Treatment B) | Treatment Sequence 5: (Treatment B + Treatment A + Treatment C) | Treatment Sequence 6: (Treatment C + Treatment B + Treatment A)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least one dose of the study drug and were included in the safety evaluations.
Groups:
- Sequence 2: (Treatment B + Treatment C + Treatment A): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 under fasting condition as Treatment A . There was a washout period of not less than 4 days between each treatment period.
- Sequence 6: (Treatment C + Treatment B + Treatment A): TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal 30 minutes after dosing as Treatment C, followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 2 administered with a high fat or high calorie meal 30 minutes prior to dosing as Treatment B, and further followed by TAK-227 50 mg, capsule, single oral dose on Day 1 of Treatment Period 3 under fasting condition as Treatment A. There will be a washout period of not less than 4 days between each treatment period.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: (Treatment A + Treatment B + Treatment C) | Sequence 2: (Treatment B + Treatment C + Treatment A) | Treatment Sequence 3: (Treatment C + Treatment A + Treatment B) | Treatment Sequence 4: (Treatment A + Treatment C + Treatment B) | Treatment Sequence 5: (Treatment B + Treatment A + Treatment C) | Sequence 6: (Treatment C + Treatment B + Treatment A) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (6.38) | 43.0 (10.23) | 39.5 (4.20) | 42.8 (8.10) | 43.0 (7.70) | 36.5 (10.47) | 42.3 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 2 | 1 | 11
  Male | 2 | 1 | 2 | 3 | 2 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 4 | 2 | 3 | 3 | 19
  Not Hispanic or Latino | 0 | 1 | 0 | 2 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1 | 2
  White | 3 | 4 | 4 | 3 | 4 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 28.613 (2.1689) | 27.055 (3.4694) | 27.795 (4.6085) | 27.640 (2.7334) | 27.380 (3.2070) | 26.280 (2.0572) | 27.460 (2.8896)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 164.5 (8.43) | 165.0 (10.03) | 162.3 (12.71) | 171.3 (11.15) | 169.8 (15.65) | 173.8 (6.65) | 167.8 (10.72)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.43 (7.135) | 74.18 (15.436) | 74.07 (18.007) | 80.78 (5.038) | 80.00 (19.588) | 79.33 (4.640) | 77.63 (11.986)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-227
Time Frame: Day 1 pre-dose and at multiple time points (up to 36 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (for example, exposure to treatment, availability of measurements, and absence of major protocol violations) were included in the PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment A: TAK-227 50 mg: TAK-227 50 mg, capsule, orally, once on Day 1 of Treatment Periods 1, 2 and 3 under fasted condition.
- Treatment B: TAK-227 50 mg: TAK-227 50 mg, capsule, orally, once on Day 1 of Treatment Periods 1, 2 and 3 with a high fat or high calorie meal 30 minutes prior to dosing.
- Treatment C: TAK-227 50 mg: TAK-227 50 mg, capsule, orally, once on Day 1 of Treatment Periods 1, 2 and 3 with a high fat or high calorie meal 30 minutes after dosing.
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
nanogram per milliliter (ng/mL) | 464.4 (89.8) | 190.9 (50.6) | 370.0 (102.6)

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-227
Time Frame: Day 1 pre-dose and at multiple time points (up to 36 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (for example, exposure to treatment, availability of measurements, and absence of major protocol violations) were included in the PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter(ng*hr/mL)
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
nanogram*hour per milliliter(ng*hr/mL) | 1582 (65.9) | 969.2 (51.2) | 1056 (53.0)

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-227
Time Frame: Day 1 pre-dose and at multiple time points (up to 36 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (for example, exposure to treatment, availability of measurements, and absence of major protocol violations) were included in the PK analyses. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter(ng*hr/mL)
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 23 | 24 | 24
nanogram*hour per milliliter(ng*hr/mL) | 1708 (52.0) | 983.7 (50.8) | 1070 (51.8)

4. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant who had signed the informed consent form (ICF) to participate in a study; it did not necessarily have to have a causal relationship with the treatment. An SAE was any untoward medical occurrence that at any dose met one or more of the following criteria: resulted in death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. A TEAE was defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From start of study drug administration up to 7 days after the last dose (up to Day 20)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants
  TEAEs | 4 | 5 | 2
  Serious TEAEs | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Based on Severity of TEAE
Description: Severity of a TEAEs were determined by following criteria: Mild: event that did not generally interfere with usual activities of daily living; Moderate: event that interfere with usual activities of daily living, causing discomfort, permanent risk of harm; Severe: AE that interrupt usual activities of daily living, significantly affects clinical status, or might require intensive therapeutic intervention.
Time Frame: From start of study drug administration up to 7 days after the last dose (up to Day 20)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Treatment B: TAK-227 50 mg: TAK-227 50 mg, capsule, orally, once on Day 1 of Periods 1, 2 and 3 with a high fat or high calorie meal 30 minutes prior to dosing.
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Mild | 3 | 5 | 2
  Moderate | 1 | 0 | 0
  Severe | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Based on Causality of TEAEs
Description: Causality of TEAEs to the study medication was assessed using the following categories: Related: An AE that followed a reasonable temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which a causal relationship was at least a reasonable possibility, that is, the relationship cannot be ruled out, although factors other than the drug, such as underlying diseases, complications, concomitant drugs and concurrent treatments, might also be responsible; Not Related: An AE that did not follow a reasonable temporal sequence from administration of a drug and/or that can reasonably be explained by other factors, such as underlying diseases, complications, concomitant medications and concurrent treatments.
Time Frame: From start of study drug administration up to 7 days after the last dose (up to Day 20)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Related TEAEs | 3 | 3 | 2
  Not Related TEAEs | 1 | 2 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs Values
Description: Vital signs included body temperature (oral or tympanic measurement), respiratory rate, blood pressure [systolic blood pressure (SBP) and diastolic blood pressure (DBP)], and pulse (beats per minute). The clinically significant change assessment was based on investigator's judgment. Number of participants with clinically significant change from baseline in vital signs values were reported.
Time Frame: Baseline to Day 13
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-Lead Electrocardiograms (ECG) Values
Description: ECGs was performed with participants in a supine position. All ECG tracings were reviewed by the investigator or designee. Number of participants with clinically significant change from baseline in ECG values were reported.
Time Frame: Baseline to Day 13
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters
Description: The clinically significant change assessment was based on investigator's judgment. Number of participants with clinically significant change from baseline in laboratory values (hematology, serum chemistry, and urinalysis) were reported.
Time Frame: Baseline to Day 13
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination
Description: Physical examination included the following body systems: (1) respiratory system; (2) cardiovascular system; (3) nervous system (4) dermatologic system; and (5) gastrointestinal system. The clinically significant change assessment was based on investigator's judgment. Number of participants with clinically significant change from baseline in physical examination values were reported.
Time Frame: Baseline to Day 13
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 7 days after the last dose (up to Day 20)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Treatment A: TAK-227 50 mg | Treatment B: TAK-227 50 mg | Treatment C: TAK-227 50 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 0/24 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: TAK-227 50 mg (N=24) | Treatment B: TAK-227 50 mg (N=24) | Treatment C: TAK-227 50 mg (N=24)
Headache (Nervous system disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT05818956/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT05818956/SAP_001.pdf